CLINICAL TRIAL: NCT03277456
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Influenza Vaccine MVA-NP+M1, Manufactured on the AGE1.CR.pIX Novel Avian Cell Line, in Healthy Adult Volunteers.
Brief Title: A Study to Determine the Safety and Immunogenicity of the Candidate Influenza Vaccine MVA-NP+M1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU008
Record Dates: First submitted 2017-09-01; First posted 2017-09-11 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Human Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single intramuscular injection of MVA-NP+M1 vaccine (Experimental): MVA-NP+M1, a novel vaccine will be administered intramuscular. The total volume given is 0.5ml and the dose given is 1.5E8 pfu. Each volunteer will receive one single injection only over a few seconds.
  Interventions: Biological: MVA-NP+M1

INTERVENTIONS:
Biological: MVA-NP+M1 — Intramuscular injection of novel vaccine

SUMMARY:
This is a first in human, phase I, open label study of the MVA viral vector (produced in the novel immortalised duck retinal cell line AGE1.CR.pIX) expressing the influenza antigens NP and M1 as a fusion protein, in healthy adult volunteers. MVA-NP+M1 will be given alone intramuscularly as a single dose.

There will be 1 study group and a total of 6 volunteers will be enrolled. Staggered enrollment will apply for the first three volunteers within the group.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-50
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
4. For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination (for women of child bearing potential only)
5. Agreement to refrain from blood donation during the course of the study
6. Provide written informed consent

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data.
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Any history of anaphylaxis in relation to vaccination
7. Pregnancy, lactation or willingness/intention to become pregnant during the study (for women of child bearing potential only)
8. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
9. History of serious psychiatric condition likely to affect participation in the study
10. Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
11. Any other serious chronic illness requiring hospital specialist supervision
12. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
13. Suspected or known injecting drug abuse in the 5 years preceding enrolment
14. Seropositive for hepatitis B surface antigen (HBsAg)
15. Seropositive for hepatitis C virus (antibodies to HCV)
16. Any clinically significant abnormal finding on screening biochemistry and haematology blood tests or urinalysis
17. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
18. Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Measure of local reactogenicity following intramuscular injection of MVA-NP+M1 | 7 days post vaccination
  Occurrence and severity of solicited local reactogenicity signs and symptoms for 7 days following vaccination using a diary card.
Measure of systemic reactogenicity following intramuscular injection of MVA-NP+M1 | 7 days post vaccination
  Occurrence and severity rating of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination using a diary card.
Measure the occurrence of adverse events following intramuscular injection of MVA-NP+M1 | 28 days post vaccination
  Occurrence and severity of unsolicited adverse events for 28 days following the vaccination using a diary card.
Assessment of safety laboratory assessments following intramuscular injection of MVA-NP+M1 | 28 days post vaccination
  Review of changes in safety laboratory measures from baseline visit to Day 2, Day 7, Day 21 and Day 28 visits
Serious Adverse Events that occur during the study | 28 days post vaccination
  Review of causality and relationship to MVA-NP+M1 for any serious adverse events during the whole study duration

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, MD, Principal Investigator — Director, The Jenner Institute, Oxford University
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No